CLINICAL TRIAL: NCT01752179
Title: The Effect of Kinesio Taping Technique on Trigger Point of Piriformis Muscle
Brief Title: Kinesio Taping Technique and Trigger Point
Acronym: KT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Welfare and Rehabilitation Science (Other)
Responsible Party: Principal Investigator, Fahimeh Hashemirad, MSc Physical therapist, University of Social Welfare and Rehabilitation Science
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90/801/T/1/5055
Record Dates: First submitted 2012-11-17; First posted 2012-12-19 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Piriformis Syndrome
Keywords: Kinesio taping; Piriformis syndrome; Trigger point
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- kinesio tape (Experimental): kinesio Tape : Width 5cm ,Length 35cm Y shape
  Interventions: Procedure: kinesio Tape : Width 5cm ,Length 35cm Y shape
- Control group (No Intervention): without using Kinesio tape

INTERVENTIONS:
Procedure: kinesio Tape : Width 5cm ,Length 35cm Y shape — In the experimental group, Kinesio taping application of piriformis according to Kenzo Kase in 2003 is modified by using unloading technique (Macdolanld, 2004). Size and Shape of Tape is Width 5cm ,Length 35cm Y shape.
  Taping method include :
  1. stretches the piriformis muscle in side lying position ,the affected leg is upper most with hip in flexion, adduction and internal rotation.
  2. puts the base of tape over the contralateral of sacrum with no tension.
  3. attaches the superior tail on the buttock over the upper part of piriformis and ends at the greater trochanter of the femur.
  4. attaches the lower tail by lifting up the soft tissue and ends at the greater trochanter of the femur.
  This is an origin to insertion application.
  Arms: kinesio tape

SUMMARY:
Kinesio taping is a novel method which recently has emerged as a viable option to treat of various musculoskeletal and neuromuscular deficits. The application of tape to injured soft tissues and joints provides support and protection for these structures. Many different techniques are used for injury prevention, treatment, rehabilitation, proprioception and sport. Elastic adhesive tape may be used to unload Myofacial Trigger Points (MTrPs), A trigger point can be located in fascia, ligaments, muscles, and tendons; however, MTrPs are also found in skeletal muscles and/or their fascia. An MTrP is a hyperirritable spot, associated with a taut band of a skeletal muscle that is painful on compression or stretch, and that can give rise to a typical referred pain pattern as well as autonomic phenomena. The use of tape along muscle to unload affected soft tissue seems to be effective in the treatment of trigger points by inhibiting overactive muscle, changing the orientation of fascia and a proprioceptive effect. The purpose of study was to determine the efficacy of Kinesio taping application on trigger point of piriformis muscle.

DETAILED DESCRIPTION:
Piriformis syndrome is a peripheral neuritis of the sciatic nerve caused by an abnormal condition of the piriformis muscle. Some investigators consider it as a form of Myofacial pain syndrome which defined as the presence of exquisite tenderness at a nodule in a palpable taut band of muscle. Trigger points are able to produce referred pain, either spontaneously or on digital compression. Although myofascial trigger points are a widely recognized phenomenon in clinical practice, there remains much to be elucidated with regards to their pathophysiology. Conservative pharmacotherapy with nonsteroidal anti-inflammatory drugs (NSAID), muscle relaxants, and physical therapy modalities such as heat therapy, cold therapy, ultrasound, electrical current and stretching were traditionally used in the treatment of trigger points.

The utilization of Kinesio taping regarding to the proposed mechanisms including 1) restoring correct muscle function by supporting weakened muscles, (2) reducing congestion by improving the flow of blood and lymphatic fluid, (3) decreasing pain by stimulating neurological system, and (4) correcting misaligned joints by retrieving muscle spasm (5) enhancing proprioception through increased stimulation to cutaneous mechanoreceptors can be helpful in restoring muscle function in patients with Myofacial trigger points . However, there are not many controlled studies that have analyzed the effects of the Kinesio taping in their treatment. Therefore, the purpose of study was to determine the efficacy of KT application as an easy and appropriate method on trigger point of piriformis muscle.

ELIGIBILITY:
Inclusion Criteria:

* Having trigger point and tenderness in piriformis muscle.
* Having at least three positive physical examination tests from FAIR, Freiberg Lasegue and Beaty test.

Exclusion Criteria:

* spinal surgery
* spinal or pelvic fracture
* disc herniation,
* facet arthropathy
* sacroiliitis
* osteoarthritis or fracture of the lower extremities
* systemic disease, such as arthritis or tuberculosis

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain intensity immediately after kinesio taping application and Change from baseline in pain intensity at three day follow-up. | Three days
  Change in pain intensity measured based on visual analogue scale at baseline, immediately after kinesio taping application and three day follow up . To measure the pain intensity in patients, a 100-mm visual analogue scale (VAS) is used. Score 0 corresponds to "no pain at all" and score 100 to "the worst imaginable pain"

SECONDARY OUTCOMES:
Change from baseline in hip internal rotation immediately after kinesio taping application and Change from baseline in hip internal rotation at three day follow-up | Three days
  Hip internal rotation is measured in the prone situation at baseline, immediately after kinesio taping application and three day follow up. Patients was asked to bent knee to 90, the axis of goniometer was placed at center of knee joint and the arms of the goniometer were aligned parallel to long axis of tibia then patient moved her leg outwardly as far as she could without allowing the pelvis movement, the stationary arm was hold in the start point while moving arm was aligned to long axis of tibia at the end range of internal rotation, this range was recorded as internal rotation of hip joint.

CONTACTS AND LOCATIONS:
Overall Officials: Fahimeh Hashemirad, MSc, Principal Investigator — Akhavan Spine Physical Therapy Center, University of Social Welfare and Rehabilitation Sciences, Tehran, Iran.; Fahimeh Hashemirad, MSc, Study Director — University of Social Welfare and Rehabilitation Sciences, Evin, Tehran, Iran.
Locations (1):
- Akhavan Spine Physical Therapy Center, University of Social Welfare and Rehabilitation Sciences, Tehran, Iran